CLINICAL TRIAL: NCT01323322
Title: Healthy Aging in Neighborhoods of Diversity Across the Life Span (HANDLS)
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: University of Maryland, Baltimore (Other); Rensselaer Polytechnic Institute (Other); Johns Hopkins University (Other); Massachusetts General Hospital (Other); University of Delaware (Other); US Department of Housing and Urban Development (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909248; 09-AG-N248
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-09-29

CONDITIONS: Diabetes; Cerebrovascular Disease; Age-Associated Decline; Cardiovascular Disease
Keywords: Socioeconomic Status; Longitudinal Study; Health Disparities; Epidemiology; Diversity; Natural History
MeSH Terms: conditions — Diabetes Mellitus; Cerebrovascular Disorders; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HANDLS: A fixed cohort as an area probability sample of Baltimore City from August 2004 through November 2009.

SUMMARY:
The Healthy Aging in Neighborhoods of Diversity across the Life Span (HANDLS) study is an interdisciplinary, community-based, prospective longitudinal epidemiologic study examining the influences of race and socioeconomic status (SES) on the development of age-related health disparities among socioeconomically diverse African Americans and whites in Baltimore. This study investigates whether health disparities develop or persist due to differences in SES, differences in race, or their interaction. HANDLS is unique because it assesses physical parameters as well as evaluating genetic, biologic, demographic, and psychosocial parameters of African American and white participants over a wide range of socioeconomic statuses, longitudinally. HANDLS also employs novel research tools, mobile medical research vehicles, in hopes of improving participation rates and retention among non-traditional research participants. The domains of the HANDLS study include: nutrition, cognition, biologic biomarkers, body composition and bone quality, physical function and performance, psychology, genomics, neighborhood environment and cardiovascular disease. Utilizing data from these study domains will facilitate an understanding of selected underlying factors of persistent black-white health disparities in overall longevity, cardiovascular disease, and cognitive decline.

HANDLS recruited a fixed cohort as an area probability sample of Baltimore City from August 2004 through November 2009 as Wave 1. HANDLS Wave 2 entitled The Association of Personality and Socioeconomic status with Health Status - An Interim Follow-up Study began in June 2006 under a separate protocol. It was designed as a follow-up telephone interview approximately 18 months after the initial examination (Wave 1) was complete. Wave 2 provided interim contact with study participants, and important interim information regarding their health. Now completed, waves 3, 4 and 5 were follow-up examinations visits to our mobile Medical Research Vehicles (MRVs). In September 2020, HANDLS initiated wave 6; telephone interviews and limited in-person visits as a COVID-centric protocol. The current protocol outlines Wave 7, the fourth follow-up examination and the participants' fifth visit to our mobile Medical Research Vehicles (MRVs). Planned as a follow-up after 3-4 years, Wave 7 consists of health examinations, questionnaires, sensory assessments (visual and olfactory), health literacy assessment, renal function assessments, environmental assessments, and for a sub-set of participants; structural MRIs, a personality inventory and an examination of sleep and cognition under separate protocols. HANDLS will resume in-person examinations with wave 7 in which we will prioritize contacting participants who were not seen in wave 5.

DETAILED DESCRIPTION:
The Healthy Aging in Neighborhoods of Diversity across the Life Span (HANDLS) study is an interdisciplinary, community-based, prospective longitudinal epidemiologic study examining the influences of race and socioeconomic status (SES) on the development of age-related health disparities among socioeconomically diverse African Americans and whites in Baltimore. This study investigates whether health disparities develop or persist due to differences in SES, differences in race, or their interaction. HANDLS is unique because it assesses physical parameters as well as evaluating genetic, biologic, demographic, and psychosocial parameters of African American and white participants over a wide range of socioeconomic statuses, longitudinally. HANDLS also employs novel research tools, mobile medical research vehicles, in hopes of improving participation rates and retention among non-traditional research participants. The domains of the HANDLS study include: nutrition, cognition, biologic biomarkers, body composition and bone quality, physical function and performance, psychology, genomics, neighborhood environment and cardiovascular disease. Utilizing data from these study domains will facilitate an understanding of selected underlying factors of persistent black-white health disparities in overall longevity, cardiovascular disease, and cognitive decline.

HANDLS recruited a fixed cohort as an area probability sample of Baltimore City from August 2004 through November 2009 as Wave 1. HANDLS Wave 2 entitled The Association of Personality and Socioeconomic status with Health Status An Interim Follow-up Study began in June 2006 under a separate protocol. It was designed as a follow-up telephone interview approximately 18 months after the initial examination (Wave 1) was complete. Wave 2 provided interim contact with study participants, and important interim information regarding their health. Now completed, waves 3, 4 and 5 were follow-up examinations visits to our mobile Medical Research Vehicles (MRVs). In September 2020, HANDLS initiated wave 6; telephone interviews and limited in-person visits as a COVID-centric protocol. The current protocol outlines Wave 7, the fourth follow-up examination and the participants fifth visit to our mobile Medical Research Vehicles (MRVs). Planned as a follow-up after 3-4 years, Wave 7 consists of health examinations, questionnaires, sensory assessments (visual and olfactory), health literacy assessment, renal function assessments, environmental assessments, and for a sub-set of participants; structural MRIs, a personality inventory and an examination of sleep and cognition under separate protocols. HANDLS will resume in-person examinations with wave 7 in which we will prioritize contacting participants who were not seen in wave 5.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Verified HANDLS participants (age 30-64 at baseline recruitment)
* Able to give informed consent (or have a legal designee); and
* Must have valid picture identification.

EXCLUSION CRITERIA:

* Pregnancy
* Current cancer chemotherapy or radiation therapy
* Positive COVID test at point of care testing on examination visit date.

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The baseline HANDLS sample consists of 3720 community-dwelling African American and white adults aged 30-64. Participants were drawn from 13 neighborhoods (groups of contiguous census tracts) in Baltimore City, sampling representatively across a wide range of socioeconomic and income circumstances.
Sampling Method: Probability Sample
Enrollment: 3720 (Actual)
Dates: Start 2009-07-01 (Actual)

PRIMARY OUTCOMES:
To disentangle the relationship between race, SES, and health outcomes. | 4 to 5 years
  Health Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Michele K Evans, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is ongoing discussion within the NIA IRP and a plan has not been finalized yet.

REFERENCES:
- [Derived] Evans MK, Zonderman AB. Health Equity through Clinical Research - Meeting the Challenge of Inclusion. NEJM Evid. 2023 Jun;2(6):EVIDctw2300015. doi: 10.1056/EVIDctw2300015. Epub 2023 May 23. PMID 38320133
- [Derived] Claudel SE, Shiroma EJ, Harris TB, Mode NA, Ahuja C, Zonderman AB, Evans MK, Powell-Wiley TM. Cross-Sectional Associations of Neighborhood Perception, Physical Activity, and Sedentary Time in Community-Dwelling, Socioeconomically Diverse Adults. Front Public Health. 2019 Sep 13;7:256. doi: 10.3389/fpubh.2019.00256. eCollection 2019. PMID 31572702